CLINICAL TRIAL: NCT00683800
Title: A Double-Blind, Randomized, Placebo-Controlled Study Assessing The Safety And Efficacy Of DVS SR For The Treatment Of Vasomotor Symptoms Associated With Menopause
Brief Title: Study Evaluating The Safety And Efficacy Of Desvenlafaxine Succinate For Vasomotor Symptoms In Menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3151A2-3353; B2061011
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Vasomotor Symptoms
Keywords: Menopause; Hot Flush; Hot Flash; Desvenlafaxine succinate Sustained Release
MeSH Terms: conditions — Hot Flashes | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): desvenlafaxine succinate (DVS) SR
  Interventions: Drug: desvenlafaxine succinate (DVS) SR
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: desvenlafaxine succinate (DVS) SR — Titration with 50 mg tablets once daily for 7 days, then 100mg tablets once daily from day 8 to day 365, then taper with 50 mg tablets once daily for 7 days, followed by 25 mg tablets once daily for 7 days.
  Arms: 1
Drug: Placebo — Titration with 50 mg placebo tablets once daily for 7 days, then 100mg placebo tablets once daily from day 8 to day 365, then taper with 50 mg placebo tablets once daily for 7 days, followed by 25 mg placebo tablets once daily for 7 days.
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Desvenlafaxine Succinate (DVS) Sustained Release (SR), in comparison to placebo for the treatment of Vasomotor Symptoms (VMS) in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women who seek treatment for hot flushes
* Body Mass Index (BMI) less than or equal to 34 kg/m^2

Exclusion Criteria:

* Hypersensitivity to Venlafaxine
* Myocardial infarction an/or unstable angina within 6 months of screening
* History of seizure disorder

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2186 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (106):
- United States (89):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Vista, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Brooklyn Center, Minnesota
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Jamestown, North Dakota
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Englewood, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Erie, Pennsylvania
  - Pfizer Investigational Site, Jenkintown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Hilton Head Island, South Carolina
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Watertown, South Dakota
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Midland, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Waco, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Sandy City, Utah
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Menomonee Falls, Wisconsin
- Canada (17):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Antigonish, Nova Scotia
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Gatineau, Quebec
  - Pfizer Investigational Site, L'Ancienne-Lorette, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint Romuald, Quebec
  - Pfizer Investigational Site, Saint-Janvier, Quebec
  - Pfizer Investigational Site, Shawinigan, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Derived] Archer DF, Pinkerton JV, Guico-Pabia CJ, Hwang E, Cheng RF; Study 3353 Investigators. Cardiovascular, cerebrovascular, and hepatic safety of desvenlafaxine for 1 year in women with vasomotor symptoms associated with menopause. Menopause. 2013 Jan;20(1):47-56. doi: 10.1097/gme.0b013e3182775fe9. PMID 23266840
- [Derived] Pinkerton JV, Archer DF, Guico-Pabia CJ, Hwang E, Cheng RF. Maintenance of the efficacy of desvenlafaxine in menopausal vasomotor symptoms: a 1-year randomized controlled trial. Menopause. 2013 Jan;20(1):38-46. doi: 10.1097/GME.0b013e318274699f. PMID 23266839
- [Derived] Pinkerton JV, Constantine G, Hwang E, Cheng RF; Study 3353 Investigators. Desvenlafaxine compared with placebo for treatment of menopausal vasomotor symptoms: a 12-week, multicenter, parallel-group, randomized, double-blind, placebo-controlled efficacy trial. Menopause. 2013 Jan;20(1):28-37. doi: 10.1097/gme.0b013e31826421a8. PMID 23010882
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A2-3353&StudyName=Study%20Evaluating%20The%20Safety%20And%20Efficacy%20Of%20Desvenlafaxine%20Succinate%20For%20Vasomotor%20Symptoms%20In%20Menopausal%20Women

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3784 participants were screened, of which 1598 participants were screen failures and 2186 participants were randomly assigned to treatment.
Groups:
- DVS SR 100 mg: Desvenlafaxine Succinate Sustained Release (DVS SR) 100 milligram (mg) tablets daily until Day 365 or early withdrawal.
- Placebo: Matching placebo tablets daily until Day 365 or early withdrawal.
Period: Overall Study
Arm/Group | DVS SR 100 mg | Placebo
Started | 1101 | 1085
Treated | 1066 | 1052
Completed | 669 | 719
Not Completed | 432 | 366
Not completed — Adverse Event | 195 | 102
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 57 | 44
Not completed — Other | 5 | 2
Not completed — Protocol Violation | 13 | 16
Not completed — Withdrawal by Subject | 66 | 64
Not completed — Lack of Efficacy | 61 | 104
Not completed — Randomized, not treated | 35 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DVS SR 100 mg | Placebo | Total
Number analyzed (Participants) | 1066 | 1052 | 2118
Age Continuous [Mean (Standard Deviation); unit: Years] | 53.95 (4.90) | 53.59 (4.91) | 53.77 (4.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1066 | 1052 | 2118
  Male | 0 | 0 | 0
Daily number of moderate and severe hot flushes [Mean (Standard Deviation); unit: Hot Flushes] — Average daily number of moderate and severe hot flushes was calculated as the sum of number of moderate and severe hot flushes on each day divided by number of days with data. Moderate: sensation of heat with sweating; able to continue activity; and severe: sensation of heat with sweating; causing cessation of activity. Participants analysed were 184 and 181 for DVS SR 100 mg group and placebo group, respectively.
  Hot Flushes | 11.67 (5.62) | 11.91 (5.71) | 11.79 (5.66)
Daily severity score of hot flushes [Mean (Standard Deviation); unit: Units on a scale] — Severity: mild (sensation of heat without sweating); moderate (sensation of heat with sweating; able to continue activity) to severe (sensation of heat with sweating; causing cessation of activity). Average daily severity of hot flushes for each time period was calculated as (1*Number of mild+2*Number of moderate+3*Number of severe)/(Total number of hot flushes). For days with no hot flushes, severity score was set as 0. As this was derived from count data, there was no maximum; minimum score was 0; the higher values showed worse outcomes. n=184 (DVS SR 100 mg group); n=181 (placebo group).
  Units on a scale | 2.36 (0.34) | 2.39 (0.35) | 2.37 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Daily Number of Moderate to Severe Hot Flushes at Week 4
Description: The average daily number of moderate and severe hot flushes was calculated as the sum of the number of moderate and severe hot flushes on each day divided by the number of days with data. Moderate hot flushes: sensation of heat with sweating; able to continue activity; and severe hot flushes: sensation of heat with sweating; causing cessation of activity.
Time Frame: Baseline and Week 4
Population: Modified Intent-to-Treat(MITT) population: Participants randomized into efficacy substudy; at least 1 dose of study drug, vasomotor symptoms on at least 1 day of baseline period and 1 day of on-therapy period during initial 12 weeks. Last observation carried forward (LOCF) method was used. 1 participant in each group did not have data till Week 4.
Measure: Mean (Standard Error); unit: Hot Flushes
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 183 | 180
Hot Flushes | -6.52 (0.33) | -3.64 (0.33)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; An analysis of covariance with treatment as factor and baseline value as a covariate was used to compare DVS SR 100 mg with matching placebo. The comparison was performed at significance level of p=0.05 (two sided); Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference = -2.89, 95% CI 2-sided [-3.80 to -1.98]

2. Primary Outcome: Change From Baseline in the Average Daily Number of Moderate to Severe Hot Flushes at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: MITT population included all participants who were randomized into efficacy substudy, had at least 1 dose of study drug, had vasomotor symptoms recorded on at least 1 day of baseline period and at least 1 day of on-therapy period during initial 12 weeks of therapy. Assessment was done using last observation carried forward (LOCF) method.
Measure: Mean (Standard Error); unit: Hot Flushes
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Hot Flushes | -7.31 (0.35) | -4.52 (0.35)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference = -2.79, 95% CI 2-sided [-3.77 to -1.82]

3. Primary Outcome: Change From Baseline in the Average Daily Severity of Hot Flushes at Week 4
Description: Severity ranged from mild (sensation of heat without sweating); moderate (sensation of heat with sweating; able to continue activity) to severe (sensation of heat with sweating; causing cessation of activity). The average daily severity of hot flushes for each time period was calculated as (1*Number of mild+2*Number of moderate+3*Number of severe)/(Total number of hot flushes). For the days with no hot flushes, the severity score was set as 0. As this was derived from the count data, there was no maximum; the minimum score was 0; the higher values showed worse outcomes.
Time Frame: Baseline and Week 4
Population: MITT population: All participants randomized into efficacy substudy, had at least 1 dose of study drug, had vasomotor symptoms recorded on at least 1 day of baseline period and at least 1 day of on-therapy period during initial 12 weeks of therapy. Assessment was done using LOCF method. 1 participant in each group did not have data till Week 4.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 183 | 180
Units on a Scale | -0.47 (0.04) | -0.19 (0.04)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference = -0.28, 95% CI 2-sided [-0.40 to -0.16]

4. Primary Outcome: Change From Baseline in the Average Daily Severity of Hot Flushes at Week 12
Description: as for outcome 3
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Units on a Scale | -0.59 (0.05) | -0.28 (0.05)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference = -0.31, 95% CI 2-sided [-0.44 to -0.18]

5. Primary Outcome: Number of Participants With All Adjudicated Ischemic Cardiovascular (CV) Events
Description: Adjudicated ischemic cardiovascular events were a composite of: a) Coronary Heart Disease (CHD)-related death; b) New Myocardial Infarction (MI) (non-procedure-related MI); c) Documented new onset of unstable angina requiring hospitalization; d) Unscheduled coronary revascularization procedures (percutaneous coronary intervention) or bypass grafting.
Time Frame: Baseline up to Month 12
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 1066 | 1052
Participants
  Any ischemic CV event | 0 | 1
  CHD related death | 0 | 0
  New MI | 0 | 1
  New Onset of Unstable Angina | 0 | 0
  Unscheduled Coronary Revascularization Procedures | 0 | 0
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; Excess risk of DVS SR 100 mg over placebo per 1000 woman-years of exposure, defined as the difference in the exposure adjusted rates between the treatment groups, was obtained; Test type: Superiority or Other; Wald Formula = -1.07, 90% CI 2-sided [-2.86 to 0.72] — The 90% CI for excess risk was obtained using the Wald Formula

6. Secondary Outcome: Number of Participants With a Minimal Clinically Meaningful Decrease in the Average Daily Number of Hot Flushes
Description: A mean decrease from baseline of at least 5.35 moderate to severe hot flushes at week 12 in the participants was considered clinically meaningful.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Participants | 117 | 75
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; The proportion of participants achieving a response as defined by minimal clinically important difference (MCID) at week 12 was compared between DVS and placebo treatment groups with a Cochran-Mantel-Haenszel test; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline in the Number of Moderate and Severe Hot Flushes
Description: as for outcome 1
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Percentage of participants
  Week 4 | 58.47 | 28.89
  Week 12 | 67.93 | 44.20
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; The proportion of participants achieving at least 50% hot flush reduction from baseline at 4-week was compared between DVS and placebo treatment groups with a logistic regression model with treatment as factor and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.47, 95% CI 2-sided [2.24 to 5.36]
Statistical Analysis 2: Comparison: DVS SR 100 mg vs Placebo; The proportion of participants achieving at least 50% hot flush reduction from baseline at 12-week was compared between DVS and placebo treatment groups with a logistic regression model with treatment as factor and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.75 to 4.10]

8. Secondary Outcome: Percentage of Participants With at Least 75% Reduction From Baseline in the Number of Moderate and Severe Hot Flushes
Description: as for outcome 1
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Percentage of participants
  Week 4 | 32.79 | 10.00
  Week 12 | 41.30 | 18.23
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; The proportion of participants achieving at least 75% hot flush reduction from baseline at 4-week was compared between DVS and placebo treatment groups with a logistic regression model with treatment as factor and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.39, 95% CI 2-sided [2.47 to 7.81]
Statistical Analysis 2: Comparison: DVS SR 100 mg vs Placebo; The proportion of participants achieving at least 75% hot flush reduction from baseline at 12-week was compared between DVS and placebo treatment groups with a logistic regression model with treatment as factor and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.16, 95% CI 2-sided [1.96 to 5.09]

9. Secondary Outcome: Median Time to the First Day of 3 Consecutive Days of at Least 50% Reduction in Hot Flushes
Description: Time to response was defined as the time-to-first 50% reduction in the average daily number of moderate to severe hot flushes over 3 consecutive days.
Time Frame: Week 12
Population: MITT population included all participants who were randomized into efficacy substudy, had at least 1 dose of study drug, had vasomotor symptoms recorded on at least 1 day of baseline period and at least 1 day of on-therapy period during initial 12 weeks of therapy.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Days | 13.0 [10.0 to 18.0] | 48.0 [32.0 to 64.0]
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A log-rank test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Log Rank

10. Secondary Outcome: Change From Baseline in Adjusted Means in the Number of Moderate and Severe Hot Flushes at Month 6 and Month 12
Description: The average daily number of moderate and severe hot flushes was calculated as the sum of the number of moderate and severe hot flushes on each day divided by the number of days with data. Moderate hot flushes: sensation of heat with sweating; able to continue activity; and severe hot flushes: sensation of heat with sweating; causing cessation of activity. Adjusted mean was calculated by using change from baseline as response variable, treatment as factor, and baseline as covariate using the observed cases.
Time Frame: Baseline, Month 6 and Month 12
Population: MITT participants of the efficacy sub-study population who had non-missing average daily number of moderate and severe hot flushes. The assessment was done using observed values. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time point for each group respectively.
Measure: Mean (Standard Error); unit: Hot Flushes
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Hot Flushes
  Month 6 (n= 125, 124) | -8.65 (0.37) | -6.61 (0.37)
  Month 12 (n= 112, 102) | -7.98 (0.46) | -5.17 (0.48)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; An analysis of covariance with treatment as factor and baseline value as a covariate was used to compare DVS SR 100 mg with matching placebo. The comparison was performed at significance level of p=0.05 (two sided). (At month 6); Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference = -2.04, 95% CI 2-sided [-3.07 to -1.00]
Statistical Analysis 2: Comparison: DVS SR 100 mg vs Placebo; An analysis of covariance with treatment as factor and baseline value as a covariate was used to compare DVS SR 100 mg with matching placebo. The comparison was performed at significance level of p=0.05 (two sided). (At month 12); Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference = -2.81, 95% CI 2-sided [-4.12 to -1.51]

11. Secondary Outcome: Change From Baseline in Adjusted Means in the Hot Flush Severity Score at Month 6 and Month 12
Description: Severity: mild (heat sensation without sweating); moderate (heat sensation with sweating; able to continue activity); severe (heat sensation with sweating; causing cessation of activity). Average daily severity of hot flushes= (1*Number of mild+2*Number of moderate+3*Number of severe)/(Total number of hot flushes). Days with no hot flushes: severity score=0. As it was derived from count data, there was no maximum; minimum score=0; higher values= worse outcomes. Adjusted mean: calculated using change from baseline=response variable, treatment=factor and baseline=covariate using observed cases.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 184 | 181
Units on a Scale
  Month 6 (n= 125, 124) | -0.87 (0.07) | -0.56 (0.07)
  Month 12 (n= 112, 102) | -0.78 (0.07) | -0.45 (0.08)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA; Adjusted Mean Difference = -0.31, 95% CI 2-sided [-0.51 to -0.12]
Statistical Analysis 2: Comparison: DVS SR 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.003, ANCOVA; Adjusted Mean Difference = -0.33, 95% CI 2-sided [-0.54 to -0.11]

12. Secondary Outcome: Change From Baseline in the Total Greene Climacteric Scale (GCS) Score and GCS Subscores at Week 12
Description: GCS: a 21 item evaluation of symptoms which asked participants how bothered they were with particular symptom at the moment. Each item was scored as 0 = Not at all, 1 = A little, 2 = Quite a bit, and 3 = Extremely. A total score was derived from the sum of the 21 items (range 0-63). GCS was also used to generate 6 individual scores (psychological symptoms [range 0-33], anxiety [range 0-18], depression [range 0-15], somatic symptoms [range 0-21], vasomotor symptoms [range 0-6], and sexual dysfunction [range 0-3]). A decrease in the total climacteric score indicated an improvement in symptoms.
Time Frame: Baseline and Week 12
Population: Main study efficacy population included all participants who were randomized; had at least 1 dose of study medication; and had a baseline and at least 1 on therapy Greene Climacteric Scale (GCS) assessment or at least 1 on therapy Patient Global Impression (PGI) assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 964 | 986
Units on a Scale
  Baseline: Total Score | 22.48 (0.28) | 22.04 (0.28)
  Baseline: Anxiety Scale | 6.43 (0.10) | 6.36 (0.10)
  Baseline: Depression Scale | 4.92 (0.10) | 4.84 (0.09)
  Baseline: Sexual Dysfunction Scale | 1.60 (0.03) | 1.65 (0.03)
  Baseline: Psychological Scale | 11.35 (0.18) | 11.19 (0.18)
  Baseline: Somatic Scale | 4.54 (0.11) | 4.21 (0.11)
  Baseline: Vasomotor Scale | 4.99 (0.04) | 4.99 (0.04)
  Week 12: Total Score | -9.18 (0.25) | -6.84 (0.25)
  Week 12: Anxiety Scale | -2.81 (0.09) | -2.06 (0.09)
  Week 12: Depression Scale | -2.23 (0.08) | -1.55 (0.08)
  Week 12: Sexual Dysfunction Scale | -0.41 (0.03) | -0.36 (0.03)
  Week 12: Psychological Scale | -5.04 (0.15) | -3.62 (0.15)
  Week 12: Somatic Scale | -1.24 (0.09) | -1.02 (0.09)
  Week 12: Vasomotor Scale | -2.50 (0.05) | -1.85 (0.05)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; For Week 12: Change from baseline of the GCS Total score was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -2.34, 95% CI 2-sided [-3.05 to -1.64]
Statistical Analysis 2: Comparison: DVS SR 100 mg vs Placebo; For Week 12: Change from baseline of the GCS Anxiety scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.75, 95% CI 2-sided [-0.99 to -0.51]
Statistical Analysis 3: Comparison: DVS SR 100 mg vs Placebo; For Week 12: Change from baseline of the GCS Depression scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.67, 95% CI 2-sided [-0.89 to -0.45]
Statistical Analysis 4: Comparison: DVS SR 100 mg vs Placebo; For Week 12: Change from baseline of the GCS Sexual Dysfunction scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p = 0.162, Mixed Models Analysis; Adjusted Mean Difference = -0.05, 95% CI 2-sided [-0.13 to 0.02]
Statistical Analysis 5: Comparison: DVS SR 100 mg vs Placebo; For Week 12: Change from baseline of the GCS Psychological scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 was outcome variable, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -1.42, 95% CI 2-sided [-1.84 to -1.00]
Statistical Analysis 6: Comparison: DVS SR 100 mg vs Placebo; For Week 12: Change from baseline of the GCS Somatic scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis; Adjusted Mean Difference = -0.22, 95% CI 2-sided [-0.46 to 0.01]
Statistical Analysis 7: Comparison: DVS SR 100 mg vs Placebo; For Week 12: Change from baseline of the GCS Vasomotor scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.64, 95% CI 2-sided [-0.79 to -0.50]

13. Secondary Outcome: Change From Baseline in the Total Greene Climacteric Scale (GCS) Score and GCS Subscores at Month 6
Description: as for outcome 12
Time Frame: Baseline and Month 6
Population: Main study efficacy population included all participants who were randomized; had at least 1 dose of study medication; and had a baseline and at least 1 on therapy GCS assessment or at least 1 on therapy PGI assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 796 | 836
Units on a Scale
  Total Score | -9.84 (0.25) | -7.97 (0.25)
  Anxiety Scale | -3.06 (0.09) | -2.41 (0.09)
  Depression Scale | -2.35 (0.08) | -1.77 (0.08)
  Sexual Dysfunction Scale | -0.46 (0.03) | -0.41 (0.03)
  Psychological Scale | -5.39 (0.15) | -4.15 (0.15)
  Somatic Scale | -1.49 (0.08) | -1.31 (0.08)
  Vasomotor Scale | -2.55 (0.06) | -2.14 (0.05)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; For Month 6: Change from baseline of the GCS Total score was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -1.87, 95% CI 2-sided [-2.57 to -1.18]
Statistical Analysis 2: Comparison: DVS SR 100 mg vs Placebo; For Month 6: Change from baseline of the GCS Anxiety scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.65, 95% CI 2-sided [-0.90 to -0.41]
Statistical Analysis 3: Comparison: DVS SR 100 mg vs Placebo; For Month 6: Change from baseline of the GCS Depression scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.58, 95% CI 2-sided [-0.80 to -0.37]
Statistical Analysis 4: Comparison: DVS SR 100 mg vs Placebo; For Month 6: Change from baseline of the GCS Sexual Dysfunction scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p = 0.282, Mixed Models Analysis; Adjusted Mean Difference = -0.04, 95% CI 2-sided [-0.13 to 0.04]
Statistical Analysis 5: Comparison: DVS SR 100 mg vs Placebo; For Month 6: Change from baseline of the GCS Psychological scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -1.24, 95% CI 2-sided [-1.66 to -0.82]
Statistical Analysis 6: Comparison: DVS SR 100 mg vs Placebo; For Month 6: Change from baseline of the GCS Somatic scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p = 0.140, Mixed Models Analysis; Adjusted Mean Difference = -0.17, 95% CI 2-sided [-0.41 to 0.06]
Statistical Analysis 7: Comparison: DVS SR 100 mg vs Placebo; For Month 6: Change from baseline of the GCS Vasomotor scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6, and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.41, 95% CI 2-sided [-0.56 to -0.26]

14. Secondary Outcome: Change From Baseline in the Total Greene Climacteric Scale (GCS) Score and GCS Subscores at Month 12
Description: as for outcome 12
Time Frame: Baseline and Month 12
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 673 | 718
Units on a Scale
  Total Score | -10.60 (0.26) | -8.89 (0.25)
  Anxiety Scale | -3.25 (0.09) | -2.69 (0.09)
  Depression Scale | -2.66 (0.08) | -2.04 (0.08)
  Sexual Dysfunction Scale | -0.51 (0.03) | -0.43 (0.03)
  Psychological Scale | -5.88 (0.16) | -4.70 (0.15)
  Somatic Scale | -1.63 (0.09) | -1.61 (0.08)
  Vasomotor Scale | -2.64 (0.06) | -2.19 (0.06)
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; For Month 12: Change from baseline of the GCS Total score was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6 and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -1.71, 95% CI 2-sided [-2.42 to -1.00]
Statistical Analysis 2: Comparison: DVS SR 100 mg vs Placebo; For Month 12: Change from baseline of the GCS Anxiety scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6 and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.56, 95% CI 2-sided [-0.81 to -0.30]
Statistical Analysis 3: Comparison: DVS SR 100 mg vs Placebo; For Month 12: Change from baseline of the GCS Depression scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6 and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.62, 95% CI 2-sided [-0.83 to -0.40]
Statistical Analysis 4: Comparison: DVS SR 100 mg vs Placebo; For Month 12: Change from baseline of the GCS Sexual Dysfunction scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6 and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p = 0.082, Mixed Models Analysis; Adjusted Mean Difference = -0.08, 95% CI 2-sided [-0.17 to 0.01]
Statistical Analysis 5: Comparison: DVS SR 100 mg vs Placebo; For Month 12: Change from baseline of the GCS Psychological scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6 and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -1.18, 95% CI 2-sided [-1.61 to -0.75]
Statistical Analysis 6: Comparison: DVS SR 100 mg vs Placebo; For Month 12: Change from baseline of the GCS Somatic scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6 and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p = 0.865, Mixed Models Analysis; Adjusted Mean Difference = -0.02, 95% CI 2-sided [-0.25 to 0.21]
Statistical Analysis 7: Comparison: DVS SR 100 mg vs Placebo; For Month 12: Change from baseline of the GCS Vasomotor scale subscore was analyzed using a Mixed-effects model repeated measures (MMRM), for which changes from baseline at week 12, month 6 and month 12 were outcome variables, with treatment, week, and interaction between treatment and week as fixed effects with participant as a random effect, and with the baseline score as covariate; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -0.45, 95% CI 2-sided [-0.61 to -0.29]

15. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Symptom Rating (PGI-R) for Main Study Efficacy Population at Week 12
Description: PGI-R scale was intended to assess the study participant's perception of symptoms. Participants were requested to identify the severity of their hot flush symptoms. It was a 5-scale which ranged from 1 (None) to 5 (Severe).
Time Frame: Week 12
Population: Main study efficacy population included all participants who were randomized; had at least 1 dose of study medication; and had a baseline and at least 1 on therapy GCS assessment or at least 1 on therapy PGI assessment. Assessment was done using LOCF method.
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 961 | 982
Percentage of Participants
  1= None | 8.8 | 5.0
  2= Minimal | 27.8 | 18.5
  3= Mild | 28.9 | 26.5
  4= Moderate | 24.9 | 33.8
  5= Severe | 9.6 | 16.2
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

16. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Symptom Rating (PGI-R) for Main Study Efficacy Population at Month 6
Description: as for outcome 15
Time Frame: Month 6
Population: as for outcome 15
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 963 | 986
Percentage of Participants
  1= None | 8.5 | 5.7
  2= Minimal | 32.2 | 25.5
  3= Mild | 27.3 | 23.1
  4= Moderate | 22.9 | 31.1
  5= Severe | 9.0 | 14.6
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

17. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Symptom Rating (PGI-R) for Main Study Efficacy Population at Month 12
Description: as for outcome 15
Time Frame: Month 12
Population: as for outcome 15
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 963 | 986
Percentage of Participants
  1= None | 10.1 | 7.1
  2= Minimal | 32.2 | 27.8
  3= Mild | 25.9 | 21.0
  4= Moderate | 21.6 | 29.7
  5= Severe | 10.3 | 14.4
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

18. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Symptom Rating (PGI-R) for MITT Population of Efficacy Substudy at Week 12
Description: as for outcome 15
Time Frame: Week 12
Population: MITT population: All participants randomized into efficacy substudy; at least 1 dose of study drug, vasomotor symptoms recorded on at least 1 day of baseline period and 1 day of on-therapy period during initial 12 weeks of therapy. LOCF method was used. Participants analyzed included those who were evaluated for this particular scale.
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 172 | 175
Percentage of Participants
  1= None | 8.1 | 1.7
  2= Minimal | 20.3 | 10.9
  3= Mild | 29.1 | 16.6
  4= Moderate | 24.4 | 42.9
  5= Severe | 18.0 | 28.0
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

19. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Symptom Rating (PGI-R) for MITT Population of Efficacy Substudy at Month 6
Description: as for outcome 15
Time Frame: Month 6
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 172 | 175
Percentage of Participants
  1= None | 12.2 | 2.9
  2= Minimal | 29.7 | 18.3
  3= Mild | 27.3 | 17.7
  4= Moderate | 16.9 | 34.3
  5= Severe | 14.0 | 26.9
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

20. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Symptom Rating (PGI-R) for MITT Population of Efficacy Substudy at Month 12
Description: as for outcome 15
Time Frame: Month 12
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 172 | 175
Percentage of Participants
  1= None | 9.3 | 4.0
  2= Minimal | 28.5 | 17.1
  3= Mild | 26.7 | 12.6
  4= Moderate | 18.0 | 39.4
  5= Severe | 17.4 | 26.9
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

21. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Change (PGI-C) for Main Study Efficacy Population at Week 12
Description: PGI-C score was intended to assess the study participant's perception of changes in hot flushes. It was 7-point scale which ranged from 1 (Very Much Improved) to 7 (Very Much Worse).
Time Frame: Week 12
Population: as for outcome 15
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 962 | 983
Percentage of Participants
  1= Very Much Improved | 25.8 | 13.1
  2= Much Improved | 32.3 | 25.5
  3= Minimally Improved | 23.3 | 25.1
  4= No Change | 11.5 | 29.3
  5= Minimally Worse | 4.1 | 4.5
  6= Much Worse | 2.2 | 1.7
  7= Very Much Worse | 0.8 | 0.7
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

22. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Change (PGI-C) for Main Study Efficacy Population at Month 6
Description: as for outcome 21
Time Frame: Month 6
Population: as for outcome 15
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 963 | 986
Percentage of Participants
  1= Very Much Improved | 28.9 | 17.1
  2= Much Improved | 32.3 | 27.7
  3= Minimally Improved | 20.5 | 20.6
  4= No Change | 11.6 | 26.2
  5= Minimally Worse | 3.5 | 5.2
  6= Much Worse | 2.1 | 2.6
  7= Very Much Worse | 1.1 | 0.6
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

23. Secondary Outcome: Percentage of Participants With Categorical Scores Based on Patient Global Impression Change (PGI-C) for Main Study Efficacy Population at Month 12
Description: as for outcome 21
Time Frame: Month 12
Population: as for outcome 15
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 963 | 986
Percentage of Participants
  1= Very Much Improved | 31.0 | 19.9
  2= Much Improved | 29.2 | 24.5
  3= Minimally Improved | 21.1 | 21.5
  4= No Change | 12.7 | 26.8
  5= Minimally Worse | 2.4 | 4.4
  6= Much Worse | 2.7 | 2.0
  7= Very Much Worse | 0.9 | 0.9
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

24. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Change (PGI-C) for MITT Population of Efficacy Substudy at Week 12
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 172 | 175
Percentage of Participants
  1= Very Much Improved | 26.7 | 7.4
  2= Much Improved | 35.5 | 22.3
  3= Minimally Improved | 17.4 | 29.7
  4= No Change | 12.8 | 34.3
  5= Minimally Worse | 2.9 | 4.6
  6= Much Worse | 3.5 | 1.7
  7= Very Much Worse | 1.2 | 0.0
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

25. Secondary Outcome: Percentage of Participants With Categorical Scores on Patient Global Impression Change (PGI-C) for MITT Population of Efficacy Substudy at Month 6
Description: as for outcome 21
Time Frame: Month 6
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 172 | 175
Percentage of Participants
  1= Very Much Improved | 34.9 | 14.9
  2= Much Improved | 32.6 | 25.7
  3= Minimally Improved | 15.7 | 23.4
  4= No Change | 11.0 | 29.7
  5= Minimally Worse | 2.3 | 4.0
  6= Much Worse | 2.9 | 2.3
  7= Very Much Worse | 0.6 | 0.0
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

26. Secondary Outcome: Percentage of Participants With Categorical Scores Based on Patient Global Impression Change (PGI-C) for MITT Population of Efficacy Substudy at Month 12
Description: as for outcome 21
Time Frame: Month 12
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 172 | 175
Percentage of Participants
  1= Very Much Improved | 37.2 | 13.7
  2= Much Improved | 24.4 | 18.3
  3= Minimally Improved | 21.5 | 25.1
  4= No Change | 10.5 | 36.0
  5= Minimally Worse | 1.2 | 5.1
  6= Much Worse | 4.1 | 1.7
  7= Very Much Worse | 1.2 | 0.0
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; A Cochran-Mantel-Haenszel row mean score test was used to compare the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

27. Other Pre Specified Outcome: Number of Participants With Adjudicated Cerebrovascular Events - Any Stroke
Description: Adjudicated cerebrovascular events were identified using Standardized MedDRA Query (SMQ), for "central nervous system haemorrhages and cerebrovascular conditions". Primary assessments included: 1) definite stroke, 2) probable stroke, 3) probable transient ischemic attack (TIA), and 4) no stroke or TIA.
Time Frame: Baseline up to Month 12
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 1066 | 1052
Participants
  Any Stroke (Definite or Probable) | 1 | 0
  Definite Stroke | 0 | 0
  Probable Stroke | 1 | 0
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; Excess risk over placebo of DVS SR 100 mg per 1000 woman-years of exposure, defined as the difference in the exposure adjusted rates between the treatment groups, was obtained; Test type: Superiority or Other; Wald Formula = 1.11, 90% CI 2-sided [-0.68 to 2.9] — The 90% CI for excess risk is obtained using the Wald Formula

28. Other Pre Specified Outcome: Number of Participants With Adjudicated Cerebrovascular Events - Probable TIA
Description: as for outcome 27
Time Frame: Baseline up to Month 12
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 1066 | 1052
Participants | 1 | 0

29. Other Pre Specified Outcome: Number of Participants With Ischemic Heart Disease
Description: Potential ischaemic cardiac events were identified using the Standardized MedDRA Query (SMQ) "Ischemic Heart Disease".
Time Frame: Baseline up to Month 12
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 1066 | 1052
Participants | 4 | 2
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; Wald Formula = 2.31, 90% CI 2-sided [-2.08 to 6.71] — The 90% CI for excess risk is obtained using the Wald Formula

30. Other Pre Specified Outcome: Number of Participants With Hepatic Events
Description: Hepatic events were defined as incidence of increased Liver Function Test (AST [aspartate aminotransferase] or ALT [alanine aminotransferase]) levels greater than 5 times the ULN (upper limit of normal).
Time Frame: Baseline up to Month 12
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | DVS SR 100 mg | Placebo
Number analyzed (Participants) | 1066 | 1052
Participants | 2 | 2
Statistical Analysis 1: Comparison: DVS SR 100 mg vs Placebo; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; Wald Formula = 0.08, 90% CI 2-sided [-3.51 to 3.67] — The 90% CI for excess risk is obtained using the Wald Formula

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | DVS SR 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 43/1066 | 36/1052
Other Adverse Events (participants affected / at risk) | 941/1066 | 872/1052
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 100 mg (N=1066) | Placebo (N=1052)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Narrow anterior chamber angle (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Drug therapeutic incompatibility (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Cardiac stress test abnormal (Investigations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dermatofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ageusia (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 100 mg (N=1066) | Placebo (N=1052)
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Leukopenia (Blood and lymphatic system disorders) | 3 | 4
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic granuloma (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 2
Conduction disorder (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 35 | 33
Pulmonary valve incompetence (Cardiac disorders) | 0 | 1
Right atrial dilatation (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 7 | 7
Ventricular extrasystoles (Cardiac disorders) | 4 | 0
Keratosis follicular (Congenital, familial and genetic disorders) | 1 | 0
Mixed hyperlipidaemia (Congenital, familial and genetic disorders) | 2 | 2
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0
Conductive deafness (Ear and labyrinth disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 3 | 1
Ear canal stenosis (Ear and labyrinth disorders) | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 2 | 4
Ear disorder (Ear and labyrinth disorders) | 3 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 16 | 8
Ear pruritus (Ear and labyrinth disorders) | 1 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 2 | 0
Middle ear effusion (Ear and labyrinth disorders) | 3 | 2
Motion sickness (Ear and labyrinth disorders) | 4 | 5
Otosclerosis (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 36 | 4
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 43 | 8
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 3 | 5
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 11
Altered visual depth perception (Eye disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Asthenopia (Eye disorders) | 1 | 0
Astigmatism (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 3
Blepharospasm (Eye disorders) | 3 | 4
Cataract (Eye disorders) | 2 | 3
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 6 | 2
Dry eye (Eye disorders) | 3 | 0
Episcleritis (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 2 | 3
Eye pain (Eye disorders) | 6 | 1
Eye pruritus (Eye disorders) | 2 | 8
Eye swelling (Eye disorders) | 1 | 1
Eyelid cyst (Eye disorders) | 0 | 2
Eyelid oedema (Eye disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 2 | 0
Iritis (Eye disorders) | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 3 | 3
Macular degeneration (Eye disorders) | 1 | 1
Macular oedema (Eye disorders) | 0 | 1
Mydriasis (Eye disorders) | 6 | 1
Myopia (Eye disorders) | 0 | 1
Narrow anterior chamber angle (Eye disorders) | 1 | 0
Night blindness (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 4 | 0
Photophobia (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 1 | 0
Pinguecula (Eye disorders) | 1 | 0
Presbyopia (Eye disorders) | 1 | 0
Pupil fixed (Eye disorders) | 1 | 0
Retinal aneurysm (Eye disorders) | 1 | 1
Retinopathy hypertensive (Eye disorders) | 1 | 0
Scleral hyperaemia (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 25 | 10
Visual acuity reduced (Eye disorders) | 3 | 1
Visual impairment (Eye disorders) | 4 | 0
Vitreous degeneration (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 2 | 0
Vitreous floaters (Eye disorders) | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 22 | 20
Abdominal distension (Gastrointestinal disorders) | 16 | 8
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 23 | 24
Abdominal pain lower (Gastrointestinal disorders) | 2 | 7
Abdominal pain upper (Gastrointestinal disorders) | 39 | 41
Abdominal tenderness (Gastrointestinal disorders) | 2 | 2
Abnormal faeces (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 4 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 2 | 1
Change of bowel habit (Gastrointestinal disorders) | 2 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 118 | 40
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 79 | 56
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 88 | 15
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 63 | 50
Dysphagia (Gastrointestinal disorders) | 0 | 2
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 20 | 5
Food poisoning (Gastrointestinal disorders) | 3 | 2
Frequent bowel movements (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 4 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 20 | 18
Gingival erosion (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 2 | 3
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Gingival ulceration (Gastrointestinal disorders) | 1 | 1
Glossodynia (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 3 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 6 | 8
Hiatus hernia (Gastrointestinal disorders) | 1 | 3
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 279 | 89
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral disorder (Gastrointestinal disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 7 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 2 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1
Polyp colorectal (Gastrointestinal disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 3
Retching (Gastrointestinal disorders) | 1 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 1 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 2
Tongue dry (Gastrointestinal disorders) | 1 | 0
Tooth discolouration (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 37 | 30
Vomiting (Gastrointestinal disorders) | 50 | 26
Asthenia (General disorders) | 27 | 11
Axillary pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 9 | 11
Chest pain (General disorders) | 4 | 6
Chills (General disorders) | 28 | 8
Cyst (General disorders) | 3 | 2
Device breakage (General disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Energy increased (General disorders) | 3 | 1
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 109 | 35
Feeling abnormal (General disorders) | 6 | 3
Feeling cold (General disorders) | 2 | 2
Feeling drunk (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 3
Feeling jittery (General disorders) | 18 | 1
Feeling of body temperature change (General disorders) | 0 | 2
Generalised oedema (General disorders) | 1 | 0
Hangover (General disorders) | 2 | 0
Hunger (General disorders) | 1 | 0
Impaired healing (General disorders) | 2 | 0
Implant site reaction (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 13 | 14
Injection site haematoma (General disorders) | 1 | 0
Injection site pain (General disorders) | 2 | 2
Irritability (General disorders) | 32 | 19
Local swelling (General disorders) | 0 | 1
Malaise (General disorders) | 8 | 4
Mass (General disorders) | 0 | 2
Medical device pain (General disorders) | 0 | 1
Nodule (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 8 | 9
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 12 | 14
Pain (General disorders) | 41 | 40
Pyrexia (General disorders) | 21 | 21
Rebound effect (General disorders) | 0 | 1
Sluggishness (General disorders) | 2 | 0
Temperature intolerance (General disorders) | 1 | 1
Therapeutic response unexpected (General disorders) | 1 | 0
Thirst (General disorders) | 3 | 5
Ulcer (General disorders) | 0 | 1
Unevaluable event (General disorders) | 1 | 0
Vaccination site induration (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 0
Vestibulitis (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 2
Allergy to animal (Immune system disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 1
Allergy to chemicals (Immune system disorders) | 0 | 1
Allergy to plants (Immune system disorders) | 2 | 1
Allergy to vaccine (Immune system disorders) | 1 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 1
Food allergy (Immune system disorders) | 0 | 2
House dust allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 7 | 5
Sarcoidosis (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 17 | 22
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Anal fungal infection (Infections and infestations) | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 3 | 0
Breast abscess (Infections and infestations) | 0 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 34 | 35
Bronchitis viral (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 2 | 2
Cervicitis (Infections and infestations) | 0 | 2
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 14 | 15
Diverticulitis (Infections and infestations) | 2 | 6
Ear infection (Infections and infestations) | 12 | 17
Ear infection viral (Infections and infestations) | 1 | 0
Eye abscess (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 9 | 4
Eye infection viral (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 5 | 1
Fungal infection (Infections and infestations) | 2 | 7
Fungal skin infection (Infections and infestations) | 2 | 1
Furuncle (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 9 | 6
Gastroenteritis viral (Infections and infestations) | 24 | 15
Gastrointestinal infection (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 6 | 1
Genital herpes (Infections and infestations) | 1 | 2
Gingival infection (Infections and infestations) | 4 | 2
H1N1 influenza (Infections and infestations) | 0 | 2
Helicobacter infection (Infections and infestations) | 3 | 3
Herpes ophthalmic (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 5 | 9
Hordeolum (Infections and infestations) | 2 | 1
Incision site infection (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 2 | 1
Infected cyst (Infections and infestations) | 1 | 1
Infected sebaceous cyst (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 60 | 61
Keratitis herpetic (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 3 | 1
Labyrinthitis (Infections and infestations) | 3 | 2
Laryngitis (Infections and infestations) | 3 | 5
Localised infection (Infections and infestations) | 2 | 5
Lower respiratory tract infection (Infections and infestations) | 3 | 7
Lung infection (Infections and infestations) | 1 | 0
Lymph gland infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 162 | 168
Neurosyphilis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 3 | 5
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 15 | 11
Oral infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 4 | 1
Paronychia (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 3
Pharyngitis streptococcal (Infections and infestations) | 6 | 6
Pneumonia (Infections and infestations) | 10 | 9
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 3 | 1
Rhinitis (Infections and infestations) | 3 | 8
Secondary syphilis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 84 | 69
Sinusitis bacterial (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 3
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 2
Tinea infection (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 3 | 1
Tonsillitis (Infections and infestations) | 3 | 0
Tooth abscess (Infections and infestations) | 16 | 12
Tooth infection (Infections and infestations) | 10 | 9
Upper respiratory tract infection (Infections and infestations) | 85 | 91
Urethritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 36 | 61
Vaginal abscess (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 4 | 3
Vaginitis bacterial (Infections and infestations) | 5 | 10
Viral infection (Infections and infestations) | 3 | 6
Viral labyrinthitis (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 8 | 7
Vulval cellulitis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 3 | 13
Vulvovaginitis trichomonal (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 8
Animal bite (Injury, poisoning and procedural complications) | 3 | 1
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 7 | 8
Arthropod sting (Injury, poisoning and procedural complications) | 6 | 6
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 2
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 25 | 8
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 3 | 4
Excoriation (Injury, poisoning and procedural complications) | 4 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 12 | 5
Foot fracture (Injury, poisoning and procedural complications) | 4 | 11
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 4 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 1
Joint injury (Injury, poisoning and procedural complications) | 6 | 5
Joint sprain (Injury, poisoning and procedural complications) | 13 | 16
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 5 | 3
Medication error (Injury, poisoning and procedural complications) | 57 | 49
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1
Muscle injury (Injury, poisoning and procedural complications) | 2 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 18 | 24
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 15 | 21
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 9
Sciatic nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 2 | 2
Skin laceration (Injury, poisoning and procedural complications) | 6 | 9
Splinter (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 3 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 4
Superficial injury of eye (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 3 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 4 | 5
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 1
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0
Venomous bite (Injury, poisoning and procedural complications) | 0 | 1
Vulva injury (Injury, poisoning and procedural complications) | 1 | 0
Whiplash injury (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 3
Wrist fracture (Injury, poisoning and procedural complications) | 3 | 2
Alanine aminotransferase increased (Investigations) | 4 | 3
Albumin urine present (Investigations) | 0 | 2
Antinuclear antibody positive (Investigations) | 0 | 1
Arthroscopy (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2
Autoantibody positive (Investigations) | 0 | 1
Biopsy breast (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 22 | 21
Blood creatine increased (Investigations) | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 3 | 2
Blood iron decreased (Investigations) | 1 | 1
Blood potassium decreased (Investigations) | 0 | 2
Blood pressure diastolic increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 43 | 23
Blood pressure systolic increased (Investigations) | 2 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 14 | 9
Blood uric acid increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 7 | 4
Body temperature increased (Investigations) | 1 | 1
Bone density decreased (Investigations) | 1 | 2
Breath sounds abnormal (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 2
Electrocardiogram PR prolongation (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram T wave amplitude decreased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 3 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 13 | 5
Heart rate irregular (Investigations) | 4 | 0
Heart sounds abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 3
Intraocular pressure increased (Investigations) | 0 | 1
Lipids increased (Investigations) | 5 | 3
Liver function test abnormal (Investigations) | 5 | 3
Low density lipoprotein increased (Investigations) | 12 | 7
Mammogram abnormal (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 1
Protein total decreased (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Smear cervix abnormal (Investigations) | 0 | 1
Thyroid function test abnormal (Investigations) | 0 | 1
Total cholesterol/HDL ratio decreased (Investigations) | 0 | 1
Tuberculin test positive (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1
Urine ketone body present (Investigations) | 1 | 1
Urine output decreased (Investigations) | 1 | 0
Very low density lipoprotein increased (Investigations) | 5 | 2
Vitamin B12 decreased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 4 | 6
Weight increased (Investigations) | 38 | 33
White blood cell count decreased (Investigations) | 1 | 0
White blood cells urine (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 34 | 8
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 1
Fluid retention (Metabolism and nutrition disorders) | 2 | 3
Food craving (Metabolism and nutrition disorders) | 2 | 2
Gout (Metabolism and nutrition disorders) | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 33 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 12 | 7
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 8 | 5
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 64 | 93
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 8
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 81 | 106
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 4
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 2
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 9 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 | 7
Ligamentitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 35 | 40
Muscle tightness (Musculoskeletal and connective tissue disorders) | 5 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 27 | 36
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 10 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 46
Neck deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 31 | 46
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 6 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 71 | 73
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 4 | 5
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 3
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 12 | 7
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 3 | 0
Aphonia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 7 | 1
Burning sensation (Nervous system disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 7 | 5
Cervical myelopathy (Nervous system disorders) | 0 | 1
Circadian rhythm sleep disorder (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 1 | 0
Clumsiness (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Crying (Nervous system disorders) | 19 | 2
Decreased vibratory sense (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 21 | 6
Dizziness (Nervous system disorders) | 207 | 64
Dizziness postural (Nervous system disorders) | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 13 | 2
Exertional headache (Nervous system disorders) | 1 | 0
Head titubation (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 332 | 262
Hemicephalalgia (Nervous system disorders) | 1 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 7 | 0
Hypoaesthesia (Nervous system disorders) | 27 | 21
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 9 | 4
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 2
Mental impairment (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 25 | 18
Migraine with aura (Nervous system disorders) | 1 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 2 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 43 | 12
Poor quality sleep (Nervous system disorders) | 5 | 0
Presyncope (Nervous system disorders) | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 2 | 2
Radicular pain (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 6 | 3
Sciatica (Nervous system disorders) | 4 | 8
Sedation (Nervous system disorders) | 3 | 0
Sinus headache (Nervous system disorders) | 45 | 35
Sleep phase rhythm disturbance (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 59 | 11
Syncope (Nervous system disorders) | 1 | 4
Tension headache (Nervous system disorders) | 8 | 9
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 22 | 6
Visual field defect (Nervous system disorders) | 1 | 3
Abnormal dreams (Psychiatric disorders) | 32 | 7
Affect lability (Psychiatric disorders) | 9 | 1
Aggression (Psychiatric disorders) | 4 | 2
Agitation (Psychiatric disorders) | 10 | 4
Anger (Psychiatric disorders) | 2 | 4
Anhedonia (Psychiatric disorders) | 2 | 0
Anorgasmia (Psychiatric disorders) | 10 | 0
Anxiety (Psychiatric disorders) | 42 | 29
Apathy (Psychiatric disorders) | 1 | 4
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 1
Bruxism (Psychiatric disorders) | 3 | 0
Change in sustained attention (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 8 | 3
Decreased interest (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 15 | 9
Depression (Psychiatric disorders) | 28 | 31
Depressive symptom (Psychiatric disorders) | 1 | 0
Derealisation (Psychiatric disorders) | 1 | 3
Disorientation (Psychiatric disorders) | 6 | 3
Dissociation (Psychiatric disorders) | 2 | 0
Disturbance in sexual arousal (Psychiatric disorders) | 2 | 0
Dysphoria (Psychiatric disorders) | 0 | 1
Emotional disorder (Psychiatric disorders) | 1 | 3
Emotional distress (Psychiatric disorders) | 2 | 0
Euphoric mood (Psychiatric disorders) | 2 | 0
Feelings of worthlessness (Psychiatric disorders) | 0 | 1
Frustration (Psychiatric disorders) | 1 | 0
Impatience (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 151 | 88
Intentional drug misuse (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 24 | 5
Logorrhoea (Psychiatric disorders) | 1 | 0
Loss of libido (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Middle insomnia (Psychiatric disorders) | 4 | 0
Mood altered (Psychiatric disorders) | 8 | 7
Mood swings (Psychiatric disorders) | 11 | 3
Nervousness (Psychiatric disorders) | 21 | 4
Nightmare (Psychiatric disorders) | 10 | 3
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1
Orgasm abnormal (Psychiatric disorders) | 3 | 0
Orgasmic sensation decreased (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 2
Post-traumatic stress disorder (Psychiatric disorders) | 2 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 5 | 5
Sleep disorder (Psychiatric disorders) | 6 | 3
Sleep talking (Psychiatric disorders) | 1 | 1
Sleep terror (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 4 | 2
Suicidal ideation (Psychiatric disorders) | 2 | 2
Tearfulness (Psychiatric disorders) | 3 | 1
Tension (Psychiatric disorders) | 1 | 2
Terminal insomnia (Psychiatric disorders) | 0 | 1
Thinking abnormal (Psychiatric disorders) | 3 | 0
Tic (Psychiatric disorders) | 1 | 0
Withdrawal syndrome (Psychiatric disorders) | 14 | 0
Bladder discomfort (Renal and urinary disorders) | 1 | 0
Bladder irritation (Renal and urinary disorders) | 1 | 0
Bladder pain (Renal and urinary disorders) | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Costovertebral angle tenderness (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 7 | 4
Haematuria (Renal and urinary disorders) | 12 | 13
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 1
Ketonuria (Renal and urinary disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 4 | 1
Nephrocalcinosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 6
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 5 | 6
Polyuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 3
Renal pain (Renal and urinary disorders) | 1 | 2
Residual urine (Renal and urinary disorders) | 1 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Trigonitis (Renal and urinary disorders) | 0 | 1
Urethral caruncle (Renal and urinary disorders) | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1
Urethral prolapse (Renal and urinary disorders) | 0 | 1
Urge incontinence (Renal and urinary disorders) | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 3 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 4 | 3
Breast calcifications (Reproductive system and breast disorders) | 0 | 4
Breast cyst (Reproductive system and breast disorders) | 1 | 2
Breast discharge (Reproductive system and breast disorders) | 1 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast dysplasia (Reproductive system and breast disorders) | 0 | 2
Breast engorgement (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 3 | 4
Breast pain (Reproductive system and breast disorders) | 6 | 7
Breast swelling (Reproductive system and breast disorders) | 0 | 2
Breast tenderness (Reproductive system and breast disorders) | 3 | 14
Cervical discharge (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 3 | 1
Cervix disorder (Reproductive system and breast disorders) | 0 | 1
Coital bleeding (Reproductive system and breast disorders) | 1 | 1
Cystocele (Reproductive system and breast disorders) | 3 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 3
Dyspareunia (Reproductive system and breast disorders) | 0 | 3
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 1
Lactation disorder (Reproductive system and breast disorders) | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 3
Metrorrhagia (Reproductive system and breast disorders) | 1 | 3
Nipple pain (Reproductive system and breast disorders) | 1 | 2
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 3 | 4
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 3 | 8
Premenstrual syndrome (Reproductive system and breast disorders) | 2 | 0
Pruritus genital (Reproductive system and breast disorders) | 2 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 2 | 0
Uterine cervix stenosis (Reproductive system and breast disorders) | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 1
Uterine pain (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 10 | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 30 | 22
Vaginal stricture (Reproductive system and breast disorders) | 0 | 1
Vulva cyst (Reproductive system and breast disorders) | 1 | 2
Vulval disorder (Reproductive system and breast disorders) | 1 | 0
Vulvar erosion (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 6 | 3
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 5
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 45
Dry throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 26 | 20
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 59 | 42
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 9
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 26 | 28
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Yawning (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 6
Acne cystic (Skin and subcutaneous tissue disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 6
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Campbell de Morgan spots (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 3 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 10 | 12
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 4
Dyshidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 30 | 8
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 2
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 3 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 27 | 14
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 13
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 33 | 25
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 2 | 1
Scar (Skin and subcutaneous tissue disorders) | 2 | 0
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 2
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 2
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 19 | 10
Yellow skin (Skin and subcutaneous tissue disorders) | 1 | 0
Ex-tobacco user (Social circumstances) | 0 | 1
Stress at work (Social circumstances) | 1 | 0
Post procedural drainage (Surgical and medical procedures) | 0 | 1
Aortic dilatation (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 2
Hot flush (Vascular disorders) | 95 | 59
Hypertension (Vascular disorders) | 37 | 33
Hypotension (Vascular disorders) | 3 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 0
Peripheral coldness (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
GCS scales were analyzed only for main study efficacy population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.